CLINICAL TRIAL: NCT00289744
Title: Long-Term Follow-up Study to Evaluate the Immune Persistence of GSK Biologicals' Combined Hepatitis A / Hepatitis B Vaccine in Healthy Children
Brief Title: Long-Term Immune Persistence of GSK Biologicals' Combined Hepatitis A & B Vaccine Injected According to a 0,6 Month Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 100561 (Y6); 100562 (Year 7) (Other: GSK); 100563 (Year 8) (Other: GSK); 100564 (Year 9) (Other: GSK); 100565 (Year 10) (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Hepatitis A; Hepatitis B; TWINRIX™ ADULT
MeSH Terms: conditions — Hepatitis B; Hepatitis A

ARMS (3):
- Twinrix Group (Experimental): Subjects who received 2 doses (at Day 0 and Month 6) of Twinrix in the primary study (208127/076)
  Interventions: Biological: TWINRIX™ ADULT
- Engerix-B Additional Dose (Adult) (Experimental): Subjects aged 16 years and above who received an additional dose of EngerixTM-B (adult dose).
  Interventions: Biological: Engerix TM
- Engerix-B Additional Dose (Pediatric) (Experimental): Subjects under the age of 16 years who received an additional dose of EngerixTM-B (pediatric dose).
  Interventions: Biological: Engerix TM

INTERVENTIONS:
Biological: TWINRIX™ ADULT — 2 doses IM injection in primary study
  Arms: Twinrix Group
Biological: Engerix TM — If a subject has become seronegative for anti-HAV antibodies or lost anti-HBs seroprotection concentrations at the long-term blood sampling time point (i.e. Years 6, 7, 8, 9 or 10), he/ she will be offered an additional vaccine dose.
  Arms: Engerix-B Additional Dose (Adult); Engerix-B Additional Dose (Pediatric)

SUMMARY:
The aim of this study is to evaluate the long-term persistence of hepatitis A and B antibodies at Years 6, 7, 8, 9 and 10 after subjects received their first two doses primary vaccination schedule of combined hepatitis A/hepatitis B vaccine.

This protocol posting deals with objectives & outcome measures of the extension phase at year 6 through to 10.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
To evaluate the long-term antibody persistence, volunteers will be bled at Years 6, 7, 8, 9 and 10 after the first vaccine dose of the primary vaccination course to determine their anti-HAV and anti-HBs antibody concentrations.

If a subject has become seronegative for anti-HAV antibodies or lost anti-HBs seroprotection concentrations at the long-term blood sampling time point (i.e. Years 6, 7, 8, 9 or 10), he/ she will be offered an additional vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in this study should have participated in the primary study with combined hepatitis A/ hepatitis B vaccine.
* Written informed consent will be obtained from each subject and/ or parent or guardian of the subject before the blood sampling visit of each year.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2004-02-16 (Actual); Primary Completion 2009-04-15 (Actual); Study Completion 2009-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects enrolled in the primary study (208127/076) were invited to come back for the long-term follow-up visits at Year 6 to 10. The enrollment in the protocol section reflects the amount of subjects who came back at year 6. At follow up timepoints less subjects came back.
Pre-assignment Details: 25 subjects lost seroprotective concentrations for anti-HBs antibodies at blood sampling time-points Years 6 to 10 and were offered an additional dose of Engerix™-B after Year 10 (additional dose phase). These subjects are presented in separate sub-groups for analysis purposes while as per study protocol, the single experimental group is Twinrix.
Groups:
- Twinrix Group: Subjects who received 2 doses (at Day 0 and Month 6) of Twinrix™ in the primary study (study 208127/076)
- Engerix-B Additional Dose (Adult): Subjects who received 2 doses (at Day 0 and Month 6) of Twinrix™ in the primary study (study 208127/076). Subjects were now 16 years and above and received an additional dose of EngerixTM-B (adult dose).
- Engerix-B Additional Dose (Pediatric): Subjects who received 2 doses (at Day 0 and Month 6) of Twinrix™ in the primary study (study 208127/076). Subjects were now under the age of 16 years and received an additional dose of EngerixTM-B (pediatric dose).
Period: Year 6 Long-term Follow-up
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 178 (Number of subjects who come back at Year 6 blood sampling time-point) | 0 | 0
Completed | 178 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Year 7 Long-term Follow-up
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 175 (Subjects who came back at Year 7 blood sampling time-point) | 0 | 0
Completed | 175 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Year 8 Long-term Follow-up
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 174 (Subjects who came back at Year 8 blood sampling time-point) | 0 | 0
Completed | 174 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Year 9 Long-term Follow-up
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 173 (Subjects who came back at Year 9 blood sampling time-point) | 0 | 0
Completed | 173 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Year 10 Long-term Follow-up
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 171 (Subjects who came back at Year 10 blood sampling time-point) | 0 | 0
Completed | 171 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Additional Dose Phase
Arm/Group | Twinrix Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Started | 0 | 19 | 6
Completed | 0 | 19 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Twinrix Group
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Time Frame: Years 6, 7, 8, 9, and 10.
Population: The analysis was performed on the long-term (LT) according to protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Twinrix Group
Number analyzed (Participants) | 142
milli-international units per milliliter
  Year 6 (n=142) | 692.3 [600.9 to 797.5]
  Year 7 (n=136): number analyzed (Participants) | 136
  Year 7 (n=136) | 753.6 [650.2 to 873.5]
  Year 8 (n=132): number analyzed (Participants) | 132
  Year 8 (n=132) | 544.4 [476.9 to 621.4]
  Year 9 (n=121): number analyzed (Participants) | 121
  Year 9 (n=121) | 479.5 [413.3 to 556.3]
  Year 10 (n=120): number analyzed (Participants) | 120
  Year 10 (n=120) | 601.6 [510.6 to 708.8]

2. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration
Time Frame: At Year 6, 7, 8, 9 and 10
Population: The analysis was performed on the long-term (LT) according to protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Twinrix Group
Number analyzed (Participants) | 142
milli-international units per milliliter
  Year 6 (n= 142) | 206.2 [149.3 to 284.8]
  Year 7 (n= 136): number analyzed (Participants) | 136
  Year 7 (n= 136) | 157.5 [113.7 to 218.4]
  Year 8 (n= 132): number analyzed (Participants) | 132
  Year 8 (n= 132) | 102.7 [74.7 to 141.1]
  Year 9 (n = 121): number analyzed (Participants) | 121
  Year 9 (n = 121) | 89.1 [64.9 to 122.5]
  Year 10 (n= 120): number analyzed (Participants) | 120
  Year 10 (n= 120) | 80.7 [58.1 to 112.0]

3. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration
Time Frame: Before and 1 month after the additional dose administration
Population: The analysis was performed on the total vaccinated cohort for the additional dose.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Number analyzed (Participants) | 19 | 6
milli-international units per milliliter
  Pre-vaccination | 10.4 [8.0 to 13.5] | 8.7 [3.3 to 23.0]
  1 month after vaccination | 1431.9 [730.2 to 2807.9] | 565.9 [163.9 to 1953.5]

4. Primary Outcome: Number of Subjects With Immune Response to the Additional Dose of Engerix™-B
Description: Immune response was defined as:
  * anti-hepatitis B surface antigen (anti-HBs) antibody concentration equal or above to 10 milli-international units per milliliter (mIU/mL) at 1 month post-challenge dose in subjects seronegative at the pre-challenge time-points
  * at least a 4-fold increase in anti-HBs antibody concentrations at 1 month post-challenge dose in subjects seropositive at the pre-challenge time-points.
Time Frame: One month after the additional dose administration
Population: The analysis was performed on the total vaccinated cohort for the additional dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Number analyzed (Participants) | 19 | 6
Participants | 19 | 6

5. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) Assessed by the Investigator as Causally Related to Primary Vaccination, Study Procedures or Lack of Vaccine Efficacy
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: At Year 6, 7, 8, 9 and 10
Population: The analysis was performed on the long-term (LT) total vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 178
Participants
  Year 6 (n= 178) | 0
  Year 7 (n= 175): number analyzed (Participants) | 175
  Year 7 (n= 175) | 0
  Year 8 (n= 174): number analyzed (Participants) | 174
  Year 8 (n= 174) | 0
  Year 9 (n= 173): number analyzed (Participants) | 173
  Year 9 (n= 173) | 0
  Year 10 (n= 171): number analyzed (Participants) | 171
  Year 10 (n= 171) | 0

6. Primary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include fatigue, fever, gastrointestinal symptoms and headache.
Time Frame: During the 4-day follow-up period after additional dose
Population: The analysis was performed on the total vaccinated cohort for the additional dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Number analyzed (Participants) | 19 | 6
Participants
  Pain | 6 | 3
  Redness | 2 | 1
  Swelling | 1 | 0
  Fatigue | 2 | 3
  Fever | 0 | 1
  Gastrointestinal symptoms | 2 | 1
  Headache | 3 | 0

7. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse event (AE) covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30-day follow-up period after additional dose
Population: The analysis was performed on the total vaccinated cohort for the additional dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Number analyzed (Participants) | 19 | 6
Participants | 1 | 1

8. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 5
Time Frame: During the 30-day follow-up period after additional dose
Population: The analysis was performed on the total vaccinated cohort for the additional dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Additional Dose (Adult) | Engerix-B Additional Dose (Pediatric)
Number analyzed (Participants) | 19 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: At each time-point of the long-term follow-up period & during the 30-day follow-up period after the additional dose. Other AEs: During the 4-day (solicited AEs) or the 30-day (unsolicited AEs) follow-up period after the additional dose.
Description: Safety results were only collected for those subjects receiving an additional vaccine dose (adult or pediatric)
Arm/Group | Engerix-B Additional Dose (Adult) | Twinrix Group | Engerix-B Additional Dose (Pediatric)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0 | 0/6
Other Adverse Events (participants affected / at risk) | 8/19 | 0/0 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Additional Dose (Adult) (N=19) | Twinrix Group (N=0) | Engerix-B Additional Dose (Pediatric) (N=6)
Pain (General disorders) | 6 | 0 | 3
Redness (General disorders) | 2 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 3
Fever (General disorders) | 0 | 0 | 1
Gastrointestinal symptoms (General disorders) | 2 | 0 | 1
Headache (General disorders) | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.